CLINICAL TRIAL: NCT04094090
Title: Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Cross-Linking in Eyes With Corneal Ectasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Goodman Eye Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PXL-2211
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Keratoconus; Pellucid Marginal Corneal Degeneration; Corneal Ectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: The study is a prospective, double-armed, randomized, single study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed, accelerated (Experimental): 4 mW, 10-15 sec on, 10-15sec off, 45 minutes of illumination Intervention: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
- Pusled, accelerated (Experimental): 8 mW, 10-15 sec on, 10-15 sec off, 22.5 minutes of illumination Intervention: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution

INTERVENTIONS:
Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution — Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea
  Other Names: Corneal crosslinking

SUMMARY:
To evaluate the safety and effectiveness of the PXL Platinum 330 system for performing corneal cross-linking (CXL) for the treatment of ectatic disorders.

DETAILED DESCRIPTION:
Patients with progressive keratoconus, pellucid marginal degeneration, or at risk for post-refractive corneal ectasia will be recruited and undergo epithelial-on corneal crosslinking with the Peschke PXL-330 system using pulsed, accelerated energy delivery. Patients will undergo monitoring for 1 year, with serial measurements of corneal topography, visual acuity, intraocular pressure, pachymetry, and visual function questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Subjects who have one or both eyes that meet criteria 1 and 1 or more of the following criteria will be considered candidates for this study:

1.10 years of age or older 2. Presence of central or inferior steepening 3. Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration 4. Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as:

1. Fleischer ring
2. Vogt's striae
3. Decentered corneal apex
4. Munson's sign
5. Apical Corneal scarring consistent with Bowman's breaks
6. Scissoring of the retinoscopic reflex
7. Crab-claw appearance on topography 5. Steepest keratometry (Kmax) value ≥ 47.20 D 6. I-S keratometry difference > 1.5 D on the Pentacam map or topography map 7. Posterior corneal elevation >16 microns 8. Thinnest corneal point >300 microns 9. Contact Lens Wearers Only:

a. Removal of contact lenses for the required period of time prior to the screening refraction: Contact Lens Type Minimum Discontinuation Time Soft or Scleral 3 days Rigid gas permeable 2 weeks

Exclusion Criteria:

All subjects meeting any of the following criteria will be excluded from this study:

1. Eyes classified as either normal or atypical normal on the severity grading scheme.
2. Corneal pachymetry at the screening exam that is <300 microns at the thinnest point in the eye(s) to be treated.
3. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

   1. History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthomeoeba, etc.)
   2. Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure.
4. Pregnancy (including plan to become pregnant) or lactation during the course of the study
5. A known sensitivity to study medications
6. Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
7. Patients with a current condition that, in the physician's opinion, would interfere with or prolong epithelial healing.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-10-19 (Actual); Primary Completion 2029-10-19 (Estimated); Study Completion 2029-10-19 (Estimated)

PRIMARY OUTCOMES:
Best-contact corrected visual acuity (BSCVA) | 3, 6, and 12 months
  Change in BSCVA compared to baseline.

SECONDARY OUTCOMES:
Uncorrected visual acuity | 3, 6, and 12 months
  Change in UCVA compared to baseline.
Keratometry | 1 year
  Change in Kmax, compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Goodman Eye Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be held in a secure location. While summary outcomes data will be provided on request to other researchers and periodically at scientific conferences, protected health information will not.

DOCUMENTS (1):
  • Study Protocol (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT04094090/Prot_002.pdf